CLINICAL TRIAL: NCT07049185
Title: A Single-Arm Clinical Trial of QL1706 Combined With Celecoxib in Patients With Advanced Esophageal Squamous Cell Carcinoma After Prior ICI Therapy
Brief Title: QL1706 Plus Celecoxib in Advanced Esophageal Squamous Cell Carcinoma
Acronym: QICE-ESCC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QL-ESCC-QIBA-3001; 2025YJZ60 (Other: Peking University Cancer Hospital)
Record Dates: First submitted 2025-06-22; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: immune Checkpoint Inhibitor; QL1706; Celecoxib; ESCC; ICI-resistant
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination Therapy Group (Experimental): QL1706 Plus Celecoxib Group
  Interventions: Drug: QL1706 Plus Celecoxib Group

INTERVENTIONS:
Drug: QL1706 Plus Celecoxib Group — QL1706 (anti-PD-1/CTLA-4 bispecific antibody) will be administered at 5 mg/kg by intravenous infusion every 3 weeks. Celecoxib 200 mg will be taken orally twice daily starting on Day 1 of each 3-week treatment cycle. Treatment continues until disease progression, intolerable toxicity, or for a maximum of 2 years.

SUMMARY:
This is a single-arm, Simon's two-stage phase II clinical trial to evaluate the efficacy and safety of QL1706 (a dual PD-1 and CTLA-4 antibody) combined with celecoxib in patients with advanced esophageal squamous cell carcinoma (ESCC) who progressed after prior immune checkpoint inhibitor therapy.

DETAILED DESCRIPTION:
The study aims to explore whether the combination of QL1706 and celecoxib can improve the objective response rate in ICI-refractory ESCC. Eligible patients will receive QL1706 (5 mg/kg IV Q3W) and celecoxib (200 mg BID orally) until disease progression, unacceptable toxicity, or up to 2 years. Safety, PFS, OS, and biomarkers such as PD-L1, HER2, IL-6, and IL-8 will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent;
2. Aged 18 to 75 years, inclusive;
3. Histologically or cytologically confirmed unresectable locally advanced or metastatic esophageal squamous cell carcinoma (ESCC);
4. Radiologically confirmed disease progression after at least 6 months of prior PD-1/PD-L1 inhibitor-based treatment;
5. At least one measurable lesion per RECIST v1.1 criteria;
6. Ability to swallow oral medication;
7. ECOG performance status of 0-1;
8. Estimated life expectancy ≥12 weeks;
9. Adequate organ function (without blood transfusion or growth factors within 14 days prior to first dose), including:

   ANC ≥ 1.5 × 10⁹/L; Platelets ≥ 100 × 10⁹/L; Hemoglobin ≥ 90 g/L; Serum albumin ≥ 30 g/L; TSH ≤ ULN; if abnormal, normal FT3/FT4 is acceptable; Total bilirubin ≤ 1.5 × ULN; ALT/AST ≤ 2.5 × ULN (≤ 5 × ULN if with liver metastases); ALP ≤ 2.5 × ULN; Serum creatinine ≤ 1.5 × ULN or CrCl ≥ 50 mL/min; INR ≤ 1.5 (if not on anticoagulation);
10. Non-sterilized women of childbearing potential and male participants with such partners must agree to use medically approved contraception during and for 3 months after study drug administration. Women must test negative for serum or urine HCG within 7 days prior to first dose and not be breastfeeding.

Exclusion Criteria：

1. Any active autoimmune disease or history of autoimmune disease (e.g., autoimmune hepatitis, interstitial pneumonia, uveitis, colitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism); exceptions: childhood asthma fully resolved without treatment or vitiligo;
2. Currently using immunosuppressive therapy or systemic corticosteroids >10 mg prednisone/day (or equivalent) within 2 weeks prior to enrollment;
3. History of severe allergic reactions to monoclonal antibodies;
4. Discontinued prior PD-1/PD-L1 therapy due to treatment-related toxicity;
5. Prior exposure to anti-CTLA-4 therapy;
6. History or evidence of interstitial lung disease or active non-infectious pneumonitis;
7. Known active tuberculosis;
8. Known CNS metastases, leptomeningeal disease, or spinal cord compression;
9. Other malignancies within 5 years (excluding cured skin basal cell carcinoma or cervical carcinoma in situ);
10. Clinically significant cardiac conditions (NYHA ≥ Class II heart failure, unstable angina, MI within 1 year, clinically significant arrhythmias requiring treatment, QTc >450 ms for males or >470 ms for females);
11. Clinically significant bleeding within 3 months before enrollment or known bleeding tendency (positive fecal occult blood must be followed by endoscopy if persistent);
12. Tumor invading major blood vessels or deemed likely to invade during the study;
13. Patients with esophagotracheal or mediastinal fistulas;
14. Clinically significant pleural/ascitic/pericardial effusion requiring drainage (if resolved and stable after drainage, enrollment is allowed);
15. Arterial or venous thrombotic events within 6 months (e.g., stroke, DVT, PE);
16. Known congenital or acquired bleeding disorders;
17. Abdominal fistula, GI perforation, or intra-abdominal abscess within 6 months;
18. Prior radiotherapy, chemotherapy, or surgery within 4 weeks prior to first study dose (except bone metastasis palliative radiotherapy); biologics within 4 weeks; targeted therapy within 5 half-lives; unresolved toxicities ≥ Grade 2 (except alopecia);
19. Active infection or unexplained fever ≥38.5℃ within 7 days prior to first dose;
20. Known immunodeficiency (e.g., HIV); active HBV (HBsAg-positive with HBV DNA ≥ 2000 IU/mL); or active HCV infection;
21. Prior dual immunotherapy with PD-1 and CTLA-4 antibodies;
22. Significant bleeding history within 1 month (e.g., GI bleeding or vasculitis);
23. Live vaccine administration within 4 weeks prior to or planned during the study;
24. Other conditions deemed by the investigator to interfere with participation or study results (e.g., substance abuse, psychiatric disorders, severe lab abnormalities, or social/family limitations).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) as assessed by RECIST v1.1 | Up to 24 weeks from first dose
  Objective Response Rate (ORR) per RECIST v1.1 at 6 months

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 1 year
  Progression-Free Survival (PFS) defined as the time from the first dose to the first documented disease progression per RECIST v1.1 or death from any cause, whichever occurs first.
Overall Survival (OS) | 1 year
  Overall Survival (OS) defined as the time from the first dose to death from any cause.
Duration of Response (DOR) | 1 year
  Duration of Response (DOR) for participants who achieve a complete response (CR) or partial response (PR), measured from the first documented response until documented disease progression per RECIST v1.1 or death.
Time to Response (TTR) | 1 year
  Time to Response (TTR) defined as the time from the first dose to the first documented objective response (CR or PR) per RECIST v1.1.
Disease Control Rate (DCR) | 1 year
  Disease Control Rate (DCR) defined as the percentage of participants achieving CR, PR, or stable disease (SD) as per RECIST v1.1.
Safety Assessment | 1 year
  Incidence and severity of adverse events as assessed by CTCAE v5.0.